CLINICAL TRIAL: NCT01795976
Title: A Phase II Trial to Assess the Activity of NY-ESO-1 Targeted T Cells in Advanced Oesophagogastric Cancer
Brief Title: NY-ESO-1 T Cells in OG Cancer
Acronym: ATTACK-OG
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawal of funding
Sponsor: Fiona Thistlethwaite (Other)
Collaborators: The Christie NHS Foundation Trust (Other); Erasmus Medical Center (Other); Ospedale San Raffaele (Other); University College London Hospitals (Other); Karolinska University Hospital (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Fiona Thistlethwaite, Consultant Medical Oncologist, The Christie NHS Foundation Trust
Organization: The Christie NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12_DOG14_22
Record Dates: First submitted 2013-01-10; First posted 2013-02-21 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Oesophageal Cancer
Keywords: Oesophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cyclophosphamide; fludarabine; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NY-ESO-1 T cells (Experimental): NY-ESO-1 T cells are T cells engineered to target the tumour antigen NY-ESO-1. Autologous T cells are obtained from eligible patients who have NY-ESO-1 positive tumours and who are Human Leukocyte Antigen serotype "A" serotype group (HLA2) positive. The T cells undergo lentiviral transduction with NY-ESO-1 specific nucleic acid under Good Manufacturing Practice (GMP) conditions. The patient will then undergo preconditioning chemotherapy with a regime of cyclophosphamide 60mg/kg/day day -7 and -6 followed by fludarabine 25mg/m2 day -5 to -1. They will receive autologous NY-ESO-1 T cells on day 0 and following on from that they will receive up to 14 doses of intravenous IL-2 at a dose of 100000 units per kg..
  Interventions: Genetic: NY-ESO-1 T cells; Drug: cyclophosphamide; Drug: Fludarabine; Biological: Interleukin 2

INTERVENTIONS:
Genetic: NY-ESO-1 T cells
Drug: cyclophosphamide — cyclophosphamide 60mg/kg/day day -7 and day -6
Drug: Fludarabine — Fludarabine given 25mg/m2 day -5 to day -1
Biological: Interleukin 2 — Interleukin 2 (IL2) immunotherapy given day 0 to day 6
  Other Names: IL2

SUMMARY:
This is a trial of adoptive T cell therapy using the patient's own T cells, genetically engineered to target the tumour associated antigen NY-ESO-1 (New York esophageal squamous cell carcinoma 1). Eligible patients will undergo leukapheresis (a process to remove white blood cells) to retrieve sufficient T cells which will be gene modified and expanded in the laboratory. Patients will undergo preconditioning chemotherapy with cyclophosphamide (60mg/kg) day -7 and day -6, followed by fludarabine (25mg/m2) day -5 to day -1. The NY-ESO-1 gene modified cells will be re-infused on day 0 and the patients will receive up to 14 doses of intravenous Interleukin2 (100000 U/kg) from day 0 to day 4.

The primary objective of response rate according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria will be assessed by CT scans carried out at week 6, week 12 and at 12 weekly intervals thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed oesophagogastric cancer with confirmed evidence of metastatic disease and to have failed or refused standard therapies.
* There must be measurable disease
* Patients may have had any previous systemic therapies provided they are otherwise fit for treatment
* Age equal to or greater than 18 years
* World Health Organisation (WHO) performance status of 0 or 1
* Patients must be HLA-A2 positive
* Their tumour must stain positive by immunohistochemistry for NY-ESO-1 (either diagnostic or more recent biopsy is acceptable)
* Life expectancy >3months
* Left ventricular ejection fraction (LVEF) > 50% as measured by ECHO or Multi Gated Acquisition Scan (MUGA)
* Haematological and biochemical indices:
* Haemoglobin (Hb) ≥ 8.0 g/dL
* Neutrophils ≥ 1.0 x 10*9/L
* Platelets (Plts) ≥ 100 x 10*9/L
* Any of the following abnormal baseline liver function tests:
* serum bilirubin ≤ 20 mmol/l (ULN)
* alanine aminotransferase (ALT) and/or
* aspartate aminotransferase (AST) and/or
* ≤ 3 x ULN unless patient has liver metastases when can be < 5 x ULN.
* Serum creatinine ≤ 0.15 mmol/L or creatinine clearance > 50 ml/min
* These measurements must be performed prior to leukaphereses and again prior to commencing preconditioning chemotherapy.
* The chemotherapy to be used in this trial is non-myeloablative, but where patients have had previous high dose chemotherapy, an autologous haemopoietic stem cell backup harvest, for stem cell rescue, will be obtained prior to commencing therapy in this trial. Similarly, where there is concern about a patient's bone marrow reserves, for example due to multiple previous lines of myelosuppressive chemotherapy a backup stem cell harvest should also be obtained.
* Female patients of child-bearing potential must have a negative serum or urine pregnancy test prior treatment and agree to use appropriate medically approved contraceptive precautions for four weeks prior to entering the trial, during the trial, and for six months afterwards.
* Male patients must agree to use barrier method contraception during the treatment and for six months afterwards.
* Able to provide full written informed consent.

Exclusion Criteria:

* Those receiving radiotherapy, biological therapy, endocrine therapy, immunotherapy, systemic steroids, or chemotherapy during the previous four weeks (six weeks for nitrosoureas and Mitomycin-C) prior to treatment or during the course of the treatment.
* All toxic manifestations of previous treatment must have resolved. Exceptions to this are alopecia or certain Grade 1 toxicities, which an investigator considers should not exclude the patient.
* Participation in any other clinical trial within the previous 30 days or during the course of this treatment.
* Previous allogeneic transplant.
* Clinically significant cardiac disease.
* Patients who are high medical risks because of non-malignant systemic disease, including those with active infection, uncontrolled cardiac or respiratory disease, or other serious medical or psychiatric disorders which in the lead clinicians opinion would not make the patient a good candidate for adoptive T-cell therapy.
* Concurrent serious infections within the 28 days prior to treatment
* Current malignancies at other sites, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.
* Patients known or found to be serologically positive for Hepatitis B, C, HIV or Human T cell lymphotropic Virus (HTLV).
* History of systemic autoimmune disease which could be life-threatening if reactivation occurred( for example hypothyroidism would be permissible, prior rheumatoid arthritis or systemic lupus erythematosus (SLE0 would not).
* Evidence of Centra Nervous System (CNS) involvement.
* Patients who are likely to require systemic steroids or other immunosuppressive therapy.
* Pregnant and lactating women.
* Radiotherapy to >25% skeleton.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-10; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Response rate to New York esophageal squamous cell carcinoma (NYESO) T cells | 6 weeks post treatment
  To evaluate the response rate in Oesophagogastric cancer patients who are New York esophageal squamous cell carcinoma 1 (NY-ESO-1)and Human Leukocyte Antigen serotype "A" serotype group (HLA-A2) positive to adoptive cell therapy targeted to NY-ESO-1.
Response rate to NYESO T cells | 12 weeks post treatment
  To evaluate the response rate in Oesophagogastric cancer patients who are NY-ESO-1 and HLA-A2 positive to adoptive cell therapy targeted to NY-ESO-1.
Response rate to NYESO T cells | 24 weeks post treatment
  To evaluate the response rate in Oesophagogastric cancer patients who are NY-ESO-1 and HLA-A2 positive to adoptive cell therapy targeted to NY-ESO-1.
Response rate to NYESO T cells | 36 weeks post treatment
  To evaluate the response rate in Oesophagogastric cancer patients who are NY-ESO-1 and HLA-A2 positive to adoptive cell therapy targeted to NY-ESO-1.
Response rate to NYESO T cells | 48 weeks post treatment
  To evaluate the response rate in Oesophagogastric cancer patients who are NY-ESO-1 and HLA-A2 positive to adoptive cell therapy targeted to NY-ESO-1.

SECONDARY OUTCOMES:
Feasibility and tolerability of NY-ESO-1 targeted cell therapy | Feasibility will be assessed proceed to full therapy (Study day 6).
  Evaluation of feasibility and tolerability of adoptive cell therapy targeted to NY-ESO-1 in Oesophagogastric cancer patients who are NY-ESO-1 and HLA-A2 positive.
Evaluation of the progression free survival | Until progression occurs, estimated to be average of 12 months per patient.
  measuring length of time from point of cell infusion until disease progression.
Feasibility and tolerability of NY-ESO-1 targeted cell therapy | Tolerability will be assessed for follow-up period, estimated to be average of 12 months per patient.
  Evaluation of feasibility and tolerability of adoptive cell therapy targeted to NY-ESO-1 in Oesophagogastric cancer patients who are NY-ESO-1 and HLA-A2 positive.

OTHER OUTCOMES:
modified T-cell survival | 24 weeks post cell infusion
  Laboratory analysis of gene modified T-cell survival and other immunological assessments
Evaluation of Tumour marker responses. | 24 weeks post T-cell infusion
  Measuring NY-ESO levels via blood test

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom